CLINICAL TRIAL: NCT03887546
Title: Effects of a 12-week Inspiratory Muscle Training Program With Low Resistance in Patients With Multiple Sclerosis
Brief Title: Inspiratory Muscle Training in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Director, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24121989
Record Dates: First submitted 2019-01-28; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Rehabilitation; Respiration; Breathing exercise; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Respiratory Aspiration; Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Patients are assigned randomly to the two working groups, each patient only receives one of the two protocols.
Who Masked: Investigator
Masking Description: The principal investigator doesn´t know the group of the patients until the study ends.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention is administrated with Inspiratory Muscle Trainer. 20% maximum inspiratory pressure (MIP) during the first two weeks and 30% MIP after the second week.
  12 weeks, 5 days/week, 15 minutes/day.
  Interventions: Device: Inspiratory muscle trainer
- Control group (Active Comparator): Respiratory exercise program involving nasal breathing and maximum exhalation during 12 weeks, 5 days/week, 15 minutes/day
  Interventions: Procedure: Respiratory exercise

INTERVENTIONS:
Device: Inspiratory muscle trainer — The device incorporate a unidirectional valve independent of flow to guarantee constant resistance and included a specific pressure setting (in cm H2O).
  Arms: Intervention group
Procedure: Respiratory exercise — Respiratory exercise program involving nasal breathing and maximum exhalation during 12 weeks, 5 days/week, 15 minutes/day.
  Arms: Control group

SUMMARY:
Objective: To evaluate the effectiveness of a low-intensity protocol of inspiratory muscle training (IMT) to improve respiratory strength, spirometric parameters and dyspnea in patients with multiple sclerosis (MS).

Design: Clinical trial. Randomized. Participants: 67 patients with MS, distributed in two groups, intervention and control.

Intervention: Intervention group train using IMT for 12 weeks, 5 days/week, 15 minutes/day (20% maximum inspiratory pressure (MIP) during the first two weeks and 30% MIP after the second week). Control group follow a respiratory exercise program involving nasal breathing and maximum exhalation during 12 weeks, 5 days/week, 15 minutes/day.

Evaluations: Determination of the MIP and the maximum expiratory pressure (MEP); spirometry - maximum voluntary ventilation (MVV), peak expiratory flow (PEF), tidal volume (TV); dyspnea using the Borg scale and clinical evaluations.

DETAILED DESCRIPTION:
Participants:

Patients from two MS associations will be recruited to participate in a 12-week randomized trial.

The sample size calculation determine that 31 participants in each group are required to observe a minimum difference in the maximum inspiratory pressure (MIP) of 12 cm H2O, considering a power of 90%, a safety of 95% and a 10% dropout rate.

The participants in the study are diagnosed with MS, are over 18 years old, have a disability lower than 9 in the Expanded disability status scale (EDSS) and are able to understand the objectives of the study. Those participants with a current or past neurological pathology other than MS will be excluded from the study, as well as those who had had a relapse of MS or any respiratory pathology during the 4 weeks prior to the start of the study, or any other complication that may have impeded the performance of the evaluation tests or breathing techniques. All patients will be asked to carry out the 5-day weekly program at home, and a recording sheet will be provided to each participant so they will can record the time of each daily respiratory training session. All participants signed an informed consent form.

The patients will be assigned to the two groups randomly. The main researcher doesn´t meet any of the participants until the initial assessment will be carried out. The intervention group (n = 36) will receive a training protocol of IMT, while the control group (n = 31) will follow a program of nasal breathing and maximum exhalations.

Evaluation:

The participants are evaluated at the beginning and end of the intervention period.

The evaluation of MIP and MEP is performed using a pressure transducer, Elka 15, which obtains each measurement in millibar and converts it into the reference unit of centimeter of water (cm H2O) (1 mbar = 1.01973 cm H2O .), following the rules of the American thoracic society/European respiratory society (ATS / ERS) [19]. The procedure will be repeated until 3 values were obtained with a difference of less than 5%, and the highest value will be used for the analysis. The MIP of the intervention group will be assessed every 2 weeks to set the IMT workload.

Lung volumes are assessed using a datospir touch spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules will be followed [19], and the highest value of three correct measurements will be chosen. Data is collected for the following parameters: maximum voluntary ventilation (MVV), forced expiratory volume in the first second (FEV1), peak expiratory flow (PEF), mean expiratory flow (FEF25-75), vital capacity (VC), tidal volume (TV) and forced vital capacity (FVC).

Dyspnea will be measured using the modified Borg scale [20]. All evaluations will be done in the corresponding center, during the same time slot and by the same examiner for both groups.

Intervention:

For the intervention group, a protocol different from those referred to in the literature has been designed to cover the respiratory deficiencies of MS patients using IMT. The device incorporates a unidirectional valve independent of flow to guarantee constant resistance and includes a specific pressure setting (in cm H2O). During the first two weeks a MIP load of 20% will be used, followed by a load of 30% for the rest of the training period. The protocol includes 15 cycles lasting 1 minute, twice a day: one in the morning and one in the afternoon. The participants rest for 1 minute between each cycle. In total, the protocol includes 30 minutes of daily respiratory training. The patients will be instructed to inhale with enough force to reach the opening of the valve.

The training program of the control group involves nasal inhalations and maximum exhalations. The following types of breathing exercises will be carried out for 3 minutes each with a 1 minute pause for resting: abdominal breathing, chest breathing, breathing and shoulder flexion, shoulder breathing and abduction, breathing and shoulder abduction in the transverse plane. The complete protocol involves 30 minutes of daily respiratory training.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with MS
* Over 18 years old
* Disability lower than 9 in the EDSS
* Be able to understand the objectives of the study

Exclusion criteria:

* Participants with a current or past neurological pathology other than MS
* Relapse of MS or any respiratory pathology during the 4 weeks prior to the start of the study
* Any other complication that may impede the performance of the evaluation tests or breathing techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2019-04-23 (Estimated); Primary Completion 2019-07-24 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | 5 minutes
  The evaluation is performed using a pressure transducer, Elka 15, which obtainer each measurement in millibar and converted it into the reference unit of centimeter of water (cm H2O) (1 mbar = 1.01973 cm H2O), following the rules of the ATS / ERS. The procedure was repeated until 3 values were obtained with a difference of less than 5%, and the highest value was used for the analysis. The MIP of the intervention group was assessed every 2 weeks to set the IMT workload.
Maximal expiratory pressure (MEP) | 5 minutes
  The evaluation is performed using a pressure transducer, Elka 15. It is evaluated at the beginning and at the end of the interventional phase. Measure: cm H20

SECONDARY OUTCOMES:
Dyspnea | 1 minute
  Dyspnea is assessed using modified Borg scale. It is a scale between 1-10 points, 1 is the minimum and 10 is the maximum level of dyspnea or fatigue. More punctuation in the scale, more dyspnea.
Maximum voluntary ventilation (MVV) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: Liter(L) / minute(m)
Forced expiratory volume in the first second (FEV1) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Peak expiratory flow (PEF) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L / second (s)
Mean expiratory flow (FEF25-75) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L / s
Vital capacity (VC) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Tidal volume (VT) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Forced vital capacity (FVC) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L

CONTACTS AND LOCATIONS:
Overall Officials: ANA MARIA MARTIN-NOGUERAS, DR, Study Chair — University of Salamanca

IPD SHARING:
Plan to Share IPD: No